CLINICAL TRIAL: NCT05711199
Title: Effect of Glyceroltrinitrate on Human Energy Expenditure and Brown Adipose Tissue Thermogenesis
Acronym: NEXT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NEXT Study
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Brown Adipose Tissue
Keywords: energy expenditure; glyceroltrinitrate; cold exposure
MeSH Terms: interventions — Nitroglycerin

STUDY DESIGN:
Intervention Model Description: Open-label, cross-over trial in healthy volunteers with random sequence of the two study interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): 1. administration of glyceroltrinitrate (Nitroderm TTS) for 15 days.
  2. measurement of energy expenditure before and after cold exposure
  3. performing FDG-PET/CT and tissue biopsy (brown adipose tissue and muscle)
  4. measurement of glucose tolerance, triglyceride levels and energy expenditure before and after a mixed meal test.
  Interventions: Drug: Glyceroltrinitrat
- Control (No Intervention): 1. measurement of energy expenditure before and after cold exposure
  2. performing FDG-PET/CT and tissue biopsy (brown adipose tissue and muscle)
  3. measurement of glucose tolerance, triglyceride levels and energy expenditure before and after a mixed meal test.

INTERVENTIONS:
Drug: Glyceroltrinitrat — transdermal patch
  Arms: Treatment

SUMMARY:
The aim of this study is to evaluate the efficacy of glyceroltrinitrate (Nitroderm® TTS) to activate and expand human BAT as compared to mild cold exposure.

DETAILED DESCRIPTION:
The activation of brown adipose tissue in response to glyceroltrinitrate as compared to cold exposure will be studied in an open-label, cross-over trial in healthy volunteers with random sequence of the two study periods (treatment and control) seperated by a washout period of 7 days.

In the treatment phase all participants will receive Nitroderm® TTS (glyceroltrinitrate) for a total of 15 days. For better tolerability, it will be will started with a lower dose of 5mg/24h (Nitroderm® TTS) the first 5 days and after that a change to Nitroderm® TTS 10mg/24h for another 10 days will be done. Each transdermal patch will be applied for 12 hours per day (overnight) to avoid development of nitrate tolerance.

Energy expenditure will be measured by indirect calorimetry before and after a mild cold exposure by placing a medical cooling system around their midsection. Additionally brown adipose tissue activity will determined by 18F-FDG-PET/CT 30 min after injection of 75 MBq of 18F-FDG. To analyse changes in BAT and muscle which are caused by glyceroltrinitrate as compared with cold stimulus, a tissue biopsie of supraclavicular BAT and skeletal muscle (musculus vastus lateralis) will be performed.

To measure changes in glucose tolerance and triglyceride levels a mixed meal test will be performed during control and treatment phase respectively. Additionally, a indirect calorimetry will be conducted before and after mixed meal test to assess diet-induced thermogenesis, i.e. the increase in REE due to ingestion of nutrients

In control phase the same examinations will be performed, but without glyceroltrinitrat.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 to 25 kg/m2 or 30 to 35kg/m2
* Able to give informed consent as documented by signature
* Age 18 to 40 years

Exclusion Criteria:

* Contraindications to glyceroltrinitrate, e.g. known hypersensitivity or allergy
* Concomitant medication: Non-steroidal anti-inflammatory drugs (NSAID), glucocorticoids, diuretics, antihypertensives, fibrates or statins, metformin, PDE-5-inhibitors
* Clinically significant concomitant disease states (e.g. renal failure, hepatic dysfunction, cardiovascular disease, diabetes mellitus)
* Hypersensitivity to cold (e.g. Raynaud Syndrome)
* Orthostatic hypotension: systolic blood pressure decreases min. 20mmHg or diastolic blood pressure decreases min 10mmHg within 3-5min after standing up (Schellong Test at screening visit)
* History of orthostatic syncope or pre-syncope
* Blood pressure values below 100 mmHg systolic and 60 mmHg diastolic
* Allergy to local anesthetic
* Hypothyroidism without sufficient substitution
* Hyperthyroidism
* Claustrophobia
* Smoker / habitual tobacco use
* Habitual excessive alcohol use
* Weight change of >5% within 3 months prior to inclusion
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Enrolment into another study using ionizing radiation within the previous 12 months
* Pregnant or lactating women
* Lab parameters

  * Hb below lower reference limit
  * Glycated Hemoglobin (HbA1c): above 6.0%
  * Random plasma glucose >11 mM

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
BAT SUVmean | After 14 days treatment with glyceroltrinitrate or after 14 days control period respectively
  18F-FDG uptake into the supra-clavicular brown adipose tissue as determined by 18F-
BAT SUVmax | After 14 days treatment with glyceroltrinitrate or after 14 days control period respectively
  maximum SUV in supraclavicular adipose tissue (according to BARCIST 1.0)

SECONDARY OUTCOMES:
BAT Volume | After 14 days treatment with glyceroltrinitrate or after 14 days control period respectively
  volume of supraclavicular adipose tissue (according to BARCIST 1.0)
BAT glycolytic volume | After 14 days treatment with glyceroltrinitrate or after 14 days control period respectively
  volume of supraclavicular adipose tissue x SUVmean (according to BARCIST 1.0)
Energy expenditure | After 14 days treatment with glyceroltrinitrate or after 14 days control period respectively
  Quantitative change in EE above resting metabolic rate in response to the respective study intervention. Measured by indirect calorimetry.
Cold induced thermogenesis | After 14 days treatment with glyceroltrinitrate or after 14 days control period respectively
  rise in energy expenditure above baseline occurring during mild cold exposure
Mixed meal test | After 14 days treatment with glyceroltrinitrate or after 14 days control period respectively
  Changes in glucose tolerance and triglyceride levels after a mixed meal test in the respective study visit.
Skin temperature | After 14 days treatment with glyceroltrinitrate or after 14 days control period respectively
  - Changes in skin temperature and body core temperature during treatment with glyceroltrinitrate (Nitroderm® TTS) compared to control.

OTHER OUTCOMES:
Tissue biopsies of supraclavicular BAT and skeletal muscle musculus vastus lateralis | After 14 days treatment with glyceroltrinitrate or after 14 days control period respectively
  Analysis of the transcriptional changes both in BAT and muscle which are caused by the administration of glyceroltrinitrate (Nitroderm® TTS) as compared with no intervention

CONTACTS AND LOCATIONS:
Overall Officials: Matthias J Betz, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Department of Endocrinology, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No